CLINICAL TRIAL: NCT04645147
Title: Phase 1 Study of the Safety and Immunogenicity of an Epstein-Barr Virus (EBV) gp350- Ferritin Nanoparticle Vaccine in Healthy Adults With or Without EBV Infection
Brief Title: Safety and Immunogenicity of an Epstein-Barr Virus (EBV) gp350-Ferritin Nanoparticle Vaccine in Healthy Adults With or Without EBV Infection
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 210005; 21-I-0005
Record Dates: First submitted 2020-11-25; First posted 2020-11-27 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07-15

CONDITIONS: EBV; Epstein-Barr Virus Infection; Infectious Mononucleosis
Keywords: Infectious Mononucleosis; Neutralizing Antibody; CD4+ T cell response; Immune Response
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infectious Mononucleosis | interventions — Matrix-M

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EBV gp_350 Ferritin Vaccination (Experimental): Adult participants with or without prior EBV infection will receive 3 doses of vaccine
  Interventions: Biological: EBV gp350-Ferritin Vaccine; Other: Matrix-M1

INTERVENTIONS:
Biological: EBV gp350-Ferritin Vaccine — A 50 micrograms dose of EBV gp350-Ferritin vaccine will be administered intramuscularly for each vaccination at Days 0, 30, and 180 to all participants.
Other: Matrix-M1 — Each vaccine dose will consist of 50 micrograms of EBV gp350-Ferritin combined with 49 micrograms of Matrix-M1.

SUMMARY:
Background:

Epstein-Barr virus (EBV) causes most cases of infectious mononucleosis (mono). Up to 1 in 10 people who get mono can have fatigue that lasts more than 6 months. One out of 100 people can have severe complications. EBV is also associated with several types of cancer. Researchers want to test an EBV vaccine.

Objective:

To test the safety of and immune response to a new vaccine against EBV.

Eligibility:

Healthy adults ages 18-29

Design:

Participants will be screened with a medical history and physical exam. They will give a blood sample.

Screening tests will be repeated during the study.

Participants will get a dose of the study vaccine as an injection in a muscle in the upper arm. They will be observed for 30 to 60 minutes. Blood pressure, heart rate, breathing rate, and temperature will be checked. The injection site will be examined.

Participants will get a diary card. They will write down any side effects they have after the vaccine dose, or they may use an electronic diary card. Participants will be asked to write down or enter any important medical events that may occur at any time during the study.

Participants will get a vaccine dose at 2 more study visits. They will have 4 follow-up visits at different times after a vaccine dose.

Participants will have 6 telephone calls in between the in-person visits. They will also have 1 telephone call 1 year after the third dose of vaccine. If possible, this visit can occur in person.

Participation will last about 18 months. There is an optional in-person visit or telephone call 2 years after the third dose of vaccine.

DETAILED DESCRIPTION:
Study Description:

Phase 1 study to evaluate the safety and immunogenicity of a 3-dose vaccination regimen of an adjuvanted EBV gp350-Ferritin nanoparticle vaccine. Based on data reported in animal studies, our hypothesis is that this EBV vaccine will be safe and will induce a potent EBVgp350-specific immune response. Twenty EBV seropositive participants and 20 EBV seronegative participants will receive 3 doses of vaccine at 0, 1, and 6 months. Subjects will be followed until 12 months after the third dose of vaccine with an option to be followed for an additional year.

Objectives:

Primary objective:

To determine the safety and immunogenicity of an adjuvanted EBV gp350- Ferritin vaccine administered as 3 intramuscular injections to healthy adults with or without prior EBV infection.

Secondary objective: To further evaluate the immunogenicity of an adjuvanted EBV gp350-Ferritin vaccine administered to healthy adults.

Endpoints:

Primary endpoint consists of:

* Local and systemic reactogenicity signs and symptoms during the 7-day period after each vaccination
* Unsolicited adverse events up to 30 days after each vaccination
* Serious adverse events through Day 210
* Change in log10 antibody response to EBV from baseline to 1 month after the third dose of vaccine (Day 210) as measured by neutralization assay

Secondary endpoints:

* Change in log10 antibody response to EBV gp350 from baseline to Day 210 as measured by luciferase immunoprecipitation system (LIPS) assay
* Change in log10 CD4 T cell response to EBV gp350 from baseline to Day 210 as measured by intracellular cytokine staining

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. 18 to 29 years old
2. Screening procedures and evaluations performed no more than 30 days prior to scheduled administration of the first vaccine dose.
3. Ability of subject to understand and the willingness to sign a written informed consent document.
4. Stated willingness to comply with all study procedures and availability for the duration of the active phase of the study (approximately 18 months)
5. Willingness to allow storage of blood and saliva for future research.
6. In good general health as evidenced by medical history, physical examination, and laboratory screening result.
7. Subject is willing to forgo receipt of a licensed, live vaccine in the 30 days preceding each dose of vaccine or in the 30 days following each dose of vaccine. An FDA-approved inactivated, subunit or replication-defective vaccine (such as COVID-19, influenza,

   tetanus etc.) and/or a COVID-19 vaccine approved under emergency use authorization can be used >=14 days before or >=14 days after administration of the study vaccine.
8. For females of reproductive potential who are sexually active with a male partner: use of highly effective continuous contraception for at least 30 days prior to Day 0 and agreement to continue use until 60 days after the last dose of vaccine.
9. For males who are sexually active with partners of child-bearing potential: use of highly effective continuous contraception from Day 0 and agreement to continue use until 30 days after the last dose of vaccine.

   Contraceptive requirements: Because the effects of EBV gp350-Ferritin vaccine on the developing human fetus are unknown, sexually active female participants of childbearing potential must agree to use highly effective contraception as outlined below before study entry and until 60 days after the last dose of vaccine. Females of childbearing potential must have a negative pregnancy test before receiving each dose of the EBV gp350-Ferritin vaccine. During the course of the study, if a participant becomes pregnant or suspects they are pregnant, then they should inform the study staff and their primary care physician immediately. Acceptable forms of contraception are:
   * Intrauterine device (IUD) or equivalent
   * Hormonal contraceptive (e.g. consistent, timely, and continuous use of contraceptive pill, patch, ring, implant, or injection that has reached full efficacy prior to dosing). If the participant uses a contraceptive pill, path, or ring, then a barrier method (e.g. male/female condom, cap or diaphragm plus spermicide) must also be used at the time of potentially reproductive sexual activity.
   * A stable, long-term monogamous relationship with a partner who does not pose any potential pregnancy risk, e.g. has undergone a vasectomy at least 6 months prior to the first dose of vaccine or is of the same sex as the participant.
   * A hysterectomy and/or a bilateral tubal ligation or bilateral oophorectomy

   Acceptable forms of contraception for male participants include one of the following:
   * Condom plus spermicide, used before or during sexual intercourse, even if the female partner uses a contraceptive pill, patch, or ring
   * A vasectomy completed at least 6 months before the first dose of vaccine
   * Continuously and completely abstaining from sexual intercourse with a female with child-bearing potential from the first dose of vaccine until 30 days after the last dose.

   Acceptable contraception for female partners with child-bearing potential of male study participants include one of the following:
   * IUD or equivalent
   * Hormonal contraceptive (e.g. pill, patch, ring, implant or an injection used consistently and that has reached full effect prior to the first dose of vaccine)
   * Hysterectomy and/or a bilateral tubal ligation or bilateral oophorectomy

   Laboratory Criteria within 30 days or less prior to enrollment:
10. Hemoglobin within institutional normal limits or if not, then assessed and deemed not clinically significant by PI or designee
11. White blood cell (WBC) count and differential either within institutional normal reference range or if not then assessed and deemed not clinically significant by PI or designee
12. Total lymphocyte count (lymphocyte absolute) >= 800 cells/mm3 (0.8 K/mcL)
13. Platelet count equal to 125,000 - 500,000/Mm^3 (125-500 K/mcL)
14. Alanine aminotransferase (ALT) <= 1.25x upper limit of normal (ULN)
15. Serum IgG > 600 mg/dL
16. Negative human immunodeficiency virus (HIV) test.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Women who are breastfeeding or planning to become pregnant while participating through 60 days after the last dose of vaccine
2. Participant has received any of the following:

   * More than 10 days of systemic immunosuppressive medications (>=10 mg prednisone dose or its equivalent) or cytotoxic medication within the 30 days prior to first dose of vaccine or immunomodulating therapy within 180 days prior to first dose of vaccine.
   * Blood products, including immunoglobulin products, within 120 days prior to first dose of vaccine
   * Any live attenuated vaccination within 30 days prior to first dose of vaccine
   * Medically indicated subunit inactivated or replication-defective vaccines, e.g. influenza, pneumococcal, COVID-19 within 14 days of the first dose of vaccine.
   * Investigational research agents within 30 days prior to first dose or planning to receive investigational products while on study
   * Allergy treatment with antigen injections, unless on a maintenance schedule of shots no more frequently than once per month.
3. Participant has any of the following:

   * Febrile illness within 14 days of the first dose of vaccine
   * Obesity, in which any of the following are true:
   * The deltoid muscle cannot be clearly identified
   * Intramuscular (IM) vaccine administration/dosing may be compromised
   * Presence of medical comorbidities such that enrollment is not in the best interests of the participant
   * Serious reactions to vaccines
   * Hereditary, acquired, or idiopathic forms of angioedema
   * Idiopathic urticaria within the past year
   * Asthma that is not well-controlled or required emergent care, urgent care, hospitalization or intubation during the past 2 years or that requires the use of oral or intravenous steroids
   * Diabetes mellitus type 1 or type 2, excluding a history of gestational diabetes
   * Clinically significant autoimmune disease or immunodeficiency
   * Hypertension that is not well-controlled
   * Thyroid disease that is not well-controlled
   * Bleeding disorder diagnosed by doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
   * Significant bruising or bleeding difficulties with IM injections or blood draws
   * Malignancy that is active or treated malignancy for which there is no reasonable assurance of sustained cure or malignancy that is likely to recur during the study period
   * Seizure disorder other than a history of 1) febrile seizures 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the past 3 years
   * Asplenia, functional asplenia or any condition resulting in absence or removal of the spleen.
   * History of Guillain-Barre Syndrome
   * Alcohol or drug abuse or addiction
4. Any medical, psychiatric, or social condition that, in the judgement of the investigator, is a contraindication to protocol participation or impairs the participant s ability to give informed consent.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Local and systemic reactogenicity; unsolicited adverse events; serious adverse events; change in neutralizing antibody responses to EBV | Reactogenicity during the 7-day period after each dose; unsolicited adverse events up to 30 days after each dose; serious adverse events through 1 month after the third dose:; neutralizing antibody response one month after third dose
  -Local reactogenicity: pain, tenderness, redness, bruising, swelling; Systemic reactogenicity symptoms: headache, muscle pain, fatigue, chills, oral temperature, joint pain, nausea/ vomiting, diarrhea; Change in log10 antibody response to EBV from baseline to 1 month after third dose of vaccine(Day 210) as measured by neutralization assay.

SECONDARY OUTCOMES:
Change in antibody responses to EBV gp350; change in CD4+ T cell responses to EBV gp350 | Change in antibody responses and change in CD4 T cell responses at 1 month after third dose of vaccine
  -Change in log10 antibody response to EBV from baseline to 1 month after third vaccine dose measured by a luciferase immunoprecipitation assay; --Change in log10 CD4+ T cell response from baseline to one month after third dose measured by an intracellular cytokine staining assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Durkee-Shock, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will return results from CLIA approved testing done in the department of laboratory medicine to participants. Based on results and clinical judgement, we will manage and refer patients appropriately. Non-FDA approved research assay results will not be shared with patients.
Supporting Information: ICF, CSR
Time Frame: Results from the Clinical Center Laboratory will be available within one to two weeks and will be discussed by the study team.
Access Criteria: IPD will be shared with the patient. IPD will also be discussed with the study team. If collaborations are initiated the samples will be coded so that the collaborator does not know the names of the patients.

REFERENCES:
- [Background] Cohen JI, Fauci AS, Varmus H, Nabel GJ. Epstein-Barr virus: an important vaccine target for cancer prevention. Sci Transl Med. 2011 Nov 2;3(107):107fs7. doi: 10.1126/scitranslmed.3002878. PMID 22049067
- [Background] Cohen JI. Epstein-barr virus vaccines. Clin Transl Immunology. 2015 Jan 23;4(1):e32. doi: 10.1038/cti.2014.27. eCollection 2015 Jan. PMID 25671130
- [Background] Kanekiyo M, Bu W, Joyce MG, Meng G, Whittle JR, Baxa U, Yamamoto T, Narpala S, Todd JP, Rao SS, McDermott AB, Koup RA, Rossmann MG, Mascola JR, Graham BS, Cohen JI, Nabel GJ. Rational Design of an Epstein-Barr Virus Vaccine Targeting the Receptor-Binding Site. Cell. 2015 Aug 27;162(5):1090-100. doi: 10.1016/j.cell.2015.07.043. Epub 2015 Aug 13. PMID 26279189
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-I-0005.html